CLINICAL TRIAL: NCT06384391
Title: Ntestinal Ultrasound, Magnetic Resonance Enterography, and Conventional Assessment Tools Before and After Medical Treatment of Intestinal Behcet's Disease: Prospective Observational Study
Brief Title: Intestinal Ultrasound, Magnetic Resonance Enterography, and Conventional Assessment Tools Before and After Treatment of Intestinal Behcet's Disease
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-1730
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Intestinal Behcet Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The "treat-to-target" approach has recently been adopted in the treatment of inflammatory bowel disease (IBD). The basic premise is to define specific measurable targets and then adjust treatment until these targets are achieved and maintained. According to the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE)-Ⅱ statement published in 2021, the long-term treatment targets for IBD are clinical remission, endoscopic healing, absence of disability, restoration of quality of life, and normal growth in children. Symptomatic relief and normalization of serum and fecal markers were determined as short-term targets. Transmural healing in Crohn's disease and histological healing in ulcerative colitis are not formal targets but should be assessed as measures of the remission depth.

While endoscopic examination assesses the mucosal inflammatory status of the bowel wall, transmural inflammatory status needs to be evaluated with ultrasound, computed tomography (CT), or magnetic resonance enterography (MRE). Ultrasound is advantageous as it does not utilize ionizing radiation and is less costly and uncomfortable for patients, allowing more frequent use. Recent studies suggest that intestinal ultrasound is beneficial in treatment response assessment and planning in patients with Crohn's disease and ulcerative colitis. However, there is a paucity of study regarding the effectiveness of intestinal ultrasound in management of intestinal Behcet's disease. Furthermore, despite its accuracy and comprehensive imaging capabilities without radiation risk, MRE has not been widely used in the diagnosis and follow-up of the patients with intestinal Behcet's disease, and no studies have reported changes in MRE findings after treatment.

DETAILED DESCRIPTION:
Design: Prospective, single-center, cohort, observational study. Methods: The patients with intestinal Behcet's disease who have detectable bowel wall abnormality on baseline ileocolonoscopic examination, CT or MRE, and ultrasound are enrolled before starting the medical treatment. Before and until 26 weeks after the treatment, Disease Activity Index for Intestinal Behcet's disease, intestinal ultrasound, ileocolonoscopic examination, MRE, serum C-reactive protein and fecal calprotectin examinations are done.

Purpose: To investigate the accuracies of intestinal ultrasound in identifying endoscopic and clinical remissions. Additionally, to investigate the accuracies of MRE in identifying endoscopic and clinical remissions and responses. Further assessment may include cross-sectional correlation analysis between the different examination results and regression analysis to assess whether baseline examination results can predict the long-term clinical outcomes.

Sample size: 55 patients. The primary outcome of this study, the diagnostic accuracy of intestinal ultrasound in identifying endoscopic remission, has not been previous studied or reported in patients with intestinal Behcet's disease. Therefore, the investigators adopted the prospective study results published in Journal of Gastroenterology and Hepatology Open in 2020 which reported the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of intestinal ultrasound in diagnosing endoscopically active disease in Crohn disease (Sathananthan D et al. JGH Open. 2020;4(2):273-9). In that study, the sensitivity, specificity, PPV, and NPV were 91%, 83%, 91%, and 83%, respectively, in 17 patients with Crohn's disease. In the data, the accuracy must have been either 82% (14/17) or 88% (15/17). Therefore, the investigators expect the accuracy in this study to be approximately 85%. Using confidence intervals for one proportion with Score (Wilson) formula, the sample size was calculated to achieve a 95% confidence interval width of 20% for the primary outcome. This calculation resulted in a sample size of 49. Considering an expected dropout rate of 10%, the investigators aim to include a total number of 55 patients.

ELIGIBILITY:
Inclusion Criteria:

- (1) The ≥19 and <80-year-old patients who diagnosed with intestinal Behcet's disease ≥3 months ago and whose disease activity is moderate or severe.

(2) Presence of abnormality in the bowel wall detected in the endoscopic examination and CT/MRE within the period ≤3 months before enrollment

Exclusion Criteria:

* (1) Duration of intestinal Behcet's disease <3 months (2) Presence of complication that is not completely assessble with ultrasound and treating the complication is the treatment purpose (3) Absence of ultrasound finding at week 0 that correlates the abnormal findings detected in the endoscopic examination and CT/MRE (4) Suspected ulcerative colitis, Crohn's disease, unclassificed colitis, ischemic colitis, radiation proctitis, diverticular disease, or microscopic colitis (5) Evidence of active tuberculosis on chest radiograph cf. Those who were treated for ≥3 weeks for latent tuberculosis can participate in the study.

  (6) Fecal stool positive for pathogenic bacteria or Clostiridum difficile toxin.

  (7) Positive for human immunodeficient virus infection (8) Patients with hepatitis B or C or hepatic dysfunction (9) Patients who did not consent to the study participation

Ages: 19 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators are enrolling ≥19 and <80-year-old patients who were diagnosed with intestinal Behcet's disease ≥3 months ago, whose disease activity is moderate or severe, and who visit Severance Hospital to be treated. The patients with bowel wall abnormality detected in the endoscopic examination and CT/MRE within the period ≤3 months before enrollment are eligible. If there is no sonographic abnormality at week 0 that correlates the endoscopic and CT/MRE findings, the patient is not eligible. In addition, the patients who have complications not completely assessable with ultrasound and treating the complications is the treatment purpose; those who have enterocolitis attributable to the etiologies other than Behcet's disease; and those with morbidities that may affect the usual treatment of intestinal Behcet's disease are excluded.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of intestinal ultrasound in identifying endoscopic remission at 26 weeks after initiation of medical treatment | 26 weeks after initiation of the treatment.
  The accuracy is defined as (the number of the patients with both endoscopic and ultrasound remissions + number of the patients with both endoscopic and ultrasound non-remissions)/total number of the patients

SECONDARY OUTCOMES:
Accuracy of intestinal ultrasound in identifying clinical remission at 26 weeks after initiation of medical treatment | 26 weeks after initiation of the treatment.
  The accuracy is defined as (the number of the patients with both clinical and ultrasound remissions + number of the patients with both clinical and ultrasound non-remissions)/total number of the patients.
Accuracies of magnetic resonance enterography in identifying endoscopic and clinical remission at 26 weeks after initiation of medical treatment | 26 weeks after initiation of the treatment.
  1. The accuracy regarding endoscopic remission is defined as (the number of the patients with both endoscopic and magnetic resonance enterography remission + number of the patients with both endoscopic and magnetic resonance enterography non-remissions)/total number of the patients.
  2. The accuracy regarding clinical remission is defined as (the number of the patients with both clinical and magnetic resonance enterography remission + number of the patients with both clinical and magnetic resonance enterography non-remissions)/total number of the patients.
Accuracies of magnetic resonance enterography in identifying endoscopic and clinical responses at 26 weeks after initiation of medical treatment | 26 weeks after initiation of the treatment.
  1. The accuracy regarding endoscopic response is defined as (the number of the patients with both endoscopic and magnetic resonance enterography response + number of the patients with both endoscopic and magnetic resonance enterography non-response)/total number of the patients.
  2. The accuracy regarding clinical response is defined as (the number of the patients with both clinical and magnetic resonance enterography response + number of the patients with both clinical and magnetic resonance enterography non-response)/total number of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea